CLINICAL TRIAL: NCT04380805
Title: A Phase 2, Multicenter, Single Arm, Open Label Study to Evaluate the Efficacy and Safety of AK104 in Subjects With Recurrent or Metastatic Cervical Cancer
Brief Title: A Study of AK104, a PD-1/CTLA-4 Bispecific Antibody in Subjects With Recurrent/Metastatic Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: Akesobio Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-201-AU
Record Dates: First submitted 2020-05-01; First posted 2020-05-08 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Cervical Cancer; Metastatic Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AK104 (Experimental): AK104 monotherapy
  Interventions: Biological: AK104

INTERVENTIONS:
Biological: AK104 — All subjects will receive AK104 as a single agent at a dose of 6 mg/kg Q2W (Day 1 and Day 15 of each 28 day treatment cycle) via IV infusion.

SUMMARY:
This is a Phase 2, global, multicenter, open label, single arm study designed to evaluate the efficacy, safety, tolerability, pharmacokinetic (PK), and immunogenicity of AK104 monotherapy in adult subjects with previously treated recurrent or metastatic cervical carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written and signed informed consent and any locally required authorization obtained from the subject/legal representative.
2. Women aged ≥18 years at the time of study entry.
3. Subjects must have histologically or cytologically confirmed recurrent or metastatic squamous carcinoma or adenosquamous carcinoma of the cervix, and meet the following criteria: disease progression confirmed by radiologic imaging during or following prior platinum based doublet chemotherapy, with or without bevacizumab for recurrent or metastatic cervical cancer; No more than 2 prior systemic therapies in the recurrent or metastatic setting.
4. Subjects must have measurable lesions according to RECIST v1.1. The presence of measurable lesions must be confirmed by the IRRC. A previously irradiated lesion is not considered measurable and cannot be selected as a target lesion.
5. Available archived tumor tissue sample - block or a minimum of 10 unstained slides of formalin fixed paraffin embedded [FFPE] tissues - preferably from the most recent biopsy of a tumor lesion collected either at the time of or after the diagnosis of locally advanced, recurrent, and/or metastatic disease has been made.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
7. Life expectancy ≥12 weeks.
8. Adequate organ function.

Exclusion Criteria:

1. Concurrent enrollment in another clinical study, unless it is an observational (noninterventional) clinical study or the follow-up period of an interventional study.
2. Histological types of cervical cancer other than squamous carcinoma and adeno-squamous carcinoma (eg, adenocarcinoma, small cell carcinoma, clear cell carcinoma, sarcoma, etc).
3. Prior malignancy active within the previous 2 years except for the tumor for which a subject is enrolled in the study, and locally curable cancers that have been apparently cured, such as basal cell skin cancer, or carcinoma in situ of the breast.
4. Brain/central nervous system (CNS) metastases.
5. Clinically significant hydronephrosis, as determined by the investigator, not alleviated by nephrostomy or ureteral stent
6. Active infections (including tuberculosis) requiring systemic antibacterial, antifungal, or antiviral therapy within 4 weeks prior to the first dose of investigational product.
7. Known history of testing positive for human immunodeficiency virus (HIV) or known active acquired immunodeficiency syndrome.
8. Known active hepatitis B or C infections (known positive hepatitis B surface antigen [HBsAg] result or positive hepatitis C virus [HCV] antibody with detectable HCV ribonucleic acid [RNA] results).
9. Active or prior documented autoimmune disease that may relapse.
10. History of interstitial lung disease or noninfectious pneumonitis, except for those induced by radiation therapies.
11. Patients with clinically significant cardio-cerebrovascular disease.
12. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the eligibility criteria with the exception of toxicities not considered a safety risk.
13. History of severe hypersensitivity reactions to other mAbs.
14. Prior allogeneic stem cell transplantation or organ transplantation.
15. Known allergy or reaction to any component of the AK104 formulation.
16. Receipt of the following treatments or procedures: anticancer small molecule targeted agent within 2 weeks, radiation therapy within 2 weeks, other anticancer therapy within 4 weeks, any major surgery within 4 weeks, any other investigational product or procedure within 4 weeks, or agents with immunomodulatory effect within 2 weeks prior to the first dose of investigational product.
17. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily doses of prednisone or equivalent) or other immunosuppressive medications within 14 days prior to the first dose of investigational product.
18. Receipt of live attenuated vaccines within 30 days prior to the first dose of investigational product.
19. Prior exposure to any experimental antitumor vaccines, or any agent targeting T-cell costimulation or immune checkpoint pathways (eg, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, anti-CD137 or anti-OX40 antibody, etc).
20. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) assessed by Independent Radiological Review Committee (IRRC) | Up to 2 years

SECONDARY OUTCOMES:
ORR assessed by Investigator | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR per RECIST v1.1.
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Duration of Response (DoR) | Up to 2 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK104 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Number of participants with adverse events (AEs) | From the time of informed consent signed through 30 days after the last dose, up to 2 years
Minimum observed concentration (Cmin) of AK104 at steady state | From first dosing date of AK104 through 30 days post last dose of AK104, up to 2 years
Number of subjects who develop detectable anti-drug antibodies | From first dosing date of AK104 through 90 days post last dose of AK104, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Randall, MD, Study Chair — Virginia Commonwealth University
Locations (25):
- United States (19):
  - Womens Cancer Research Foundation, Newport Beach, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - BRCR Medical Center, Plantation, Florida
  - Augusta University Medical Center, Augusta, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Maryland Oncology Hematology (Plum Orchard), Silver Spring, Maryland
  - Monter Cancer Center, Lake Success, New York
  - The Blavatnik Family - Chelsea Medical Center at Mount Sinai, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Chattanooga's Program In Women's Oncology, Chattanooga, Tennessee
  - Tennessee Oncology - Centennial Clinic, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Texas Oncology-Fort Worth Cancer Center, Fort Worth, Texas
  - Lyndon B. Johnson Hospital (MD Anderson), Houston, Texas
  - Texas Oncology (Woodlands), The Woodlands, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Pacific Gynecology Specialists, P. C., Seattle, Washington
- Australia (5):
  - Monash Health, Clayton, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Ashford Cancer Centre Research, Adelaide
  - Blacktown Hospital, Blacktown
  - ICON Cancer Centre, Brisbane
- Auckland City Hospital, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No